CLINICAL TRIAL: NCT02147002
Title: Omega 3 Acids and Cardio - Vascular Complications in Patients With Chronic Kidney Disease in Stage 1-3
Brief Title: Omega-3 Acids and Cardio - Vascular Complications in Patients With Chronic Kidney Disease in Stage 1-3
Acronym: Omega-3 acids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Manitius, prof. dr hab. n.med., Collegium Medicum w Bydgoszczy
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KB305/2012; BS209 (Registry Identifier: CMBydgoszczy)
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Kidney Disease; Cardiovascular Complications
Keywords: Chronic Kidney Disease; Cardiovascular Complications
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- omega 3 acids 1 (Active Comparator): Patients with CKD stage I (GFR 90 and more ml/min/1,73 m2)
  Interventions: Dietary Supplement: Gold omega 3
- omega 3 acids 2 (Active Comparator): Patients with CKD stage II (GFR 80-89 ml/min/1,73 m2)
  Interventions: Dietary Supplement: Gold omega 3
- omega 3 acids 3 (Active Comparator): Patients with CKD stage III (GFR 30-59 ml/min/1,73 m2)
  Interventions: Dietary Supplement: Gold omega 3
- omega 3 acids 4 (Active Comparator): Patients without diabetes mellitus, hypertensions,CKD with normal level of creatinine in serum
  Interventions: Dietary Supplement: Gold omega 3

INTERVENTIONS:
Dietary Supplement: Gold omega 3 — At the beginning and at the end of the observation period, besides the clinical test, some other tests will be carried out: echocardiography, pulse wave velocity (PWV), ambulatory blood pressure monitoring (ABPM). Blood will be collected for laboratory tests such as: lipid profile, uric acid, CRP, BUN, creatinine, morphology, Ca, P, Ca x P, ionogram, xanthine oxidase, MPC1,Omega-3 acids, resolvin and protectins - the metabolites of Omega-3 acids, creatinine excretion, MPC1 excretion and excretion of uric acid.The patients will be treated with Omega-3 acids as a Gold Omega 3 preparation (2x1 capsule where 1 capsule = 1000 mg) for 6 months.
  Other Names: omega 3 acids

SUMMARY:
The National Register of Nephrology in 2007 shows, similarly to the European data, a problem of a high mortality rate among Polish dialysis patients.

The main reason of death among chronically dialysis patients are cardio - vascular system diseases. According to "The Report on the Condition of Renal Replacement Therapy in Poland in 2007", these diseases are the cause of 53% deaths in Poland. The patients with chronic kidney disease (PChN) are particularly at risk of cardio - vascular complications. These complications occur on average 30 times more often than in the whole population, and among young dialysis people, these complications occur 300 times more often. In the development of cardio - vascular complications polyunsaturated Omega-3 acids (especially eicosapentaenoic acid - EPA and docosahexaenoic acid - DHA) take a special position. The reaction of polyunsaturated Omega-3 acids on the cardiovascular system results from the enrichment of phospholipids of cell membranes within EPA and DHA. It should be noted that their impact is dependent on the type of acid and on the dose. Docosahexaenoic acid reacts with lipids and lipoproteins, blood pressure, heart rate, amount of glucose, and eicosapentaenoic acid is responsible for antiplatelet effect.

This project is aiming at defining and elaborating on the connection between Omega-3 acids, and cardiovascular complications, their influence on the functioning of the cardiovascular system, and moreover, a better understanding of the effects of therapeutic and pharmacological therapies in patients at different stages of chronic kidney disease. Carrying out this project will be a good start to shape an international project in this area.

DETAILED DESCRIPTION:
The survey will cover 90 patients from chronic kidney disease at different stages of the disease(I-III) and 30 healthy subjects as a comparison group.

At the beginning and at the end of the observation period, besides the clinical test, some other tests will be carried out: echocardiography, pulse wave velocity (PWV), ambulatory blood pressure monitoring (ABPM). Blood will be collected for laboratory tests such as: lipid profile, uric acid, C reactive protein (CRP), blood urea nitrogen (BUN), creatinine, morphology, calcium (Ca),phosphorus (P), Ca x P, ionogram, xanthine oxidase, monocyte chemoattractant protein (MPC1),Omega-3 acids, resolvin and protectins - the metabolites of Omega-3 acids, creatinine excretion, MPC1 excretion and excretion of uric acid. The patients will be treated with Omega-3 acids as a Gold Omega 3 preparation (2x1 capsule where 1 capsule = 1000 mg) for 6 months.

ELIGIBILITY:
Inclusion Criteria:

- chronic kidney disease (CKD) stage 1-3

Exclusion Criteria:

* without diabetes
* without Immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
cardiovascular complications | 6 months
  Primary measurement before the supplementation and the second measurement after 6 months of supplementation with omega-3 acid.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Manitius, prof., Study Director — Collegium Medicum in Bydgoszcz
Locations (1):
- 1Katedra i Klinika Nefrologii, Nadciśnienia Tętniczego i Chorób Wewnętrznych, Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

REFERENCES:
- [Derived] Pluta A, Strozecki P, Kesy J, Lis K, Sulikowska B, Odrowaz-Sypniewska G, Manitius J. Beneficial Effects of 6-Month Supplementation with Omega-3 Acids on Selected Inflammatory Markers in Patients with Chronic Kidney Disease Stages 1-3. Biomed Res Int. 2017;2017:1680985. doi: 10.1155/2017/1680985. Epub 2017 Nov 19. PMID 29349065